CLINICAL TRIAL: NCT02074462
Title: Managing Voriconazole Exposure During Severe Infection; Effect of Inflammation on Voriconazole Metabolic Ratio
Brief Title: Effect of Inflammation on Voriconazole Concentration
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, JWC Alffenaar, PharmD, PhD, University Medical Center Groningen
Other Study IDs: VCZ-13O30
Record Dates: First submitted 2014-02-12; First posted 2014-02-28 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Inflammation; Fungal Infection
Keywords: Voriconazole; CRP; Inflammation; Pharmacokinetics
MeSH Terms: conditions — Inflammation; Mycoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Voriconazole is a broad-spectrum antifungal agent. There is evidence for a relation between the efficacy and safety of voriconazole and voriconazole trough concentrations. There are several factors that could influence voriconazole concentrations. Inflammation could be one of these factors. In a retrospective study was observed that reduced metabolism of voriconazole was related to inflammation in patients with severe infections. Reduced metabolism of voriconazole resulted in high voriconazole levels and low N-oxide metabolite (inactive metabolite of voriconazole) levels. The purpose of this study is to determine an algorithm to guide dosing of voriconazole during severe inflammation and to develop a multiple linear regression model to describe the contribution of CRP concentrations to the variability in voriconazole levels and metabolic ratio.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 yrs
* treatment with voriconazole
* written informed consent

Exclusion Criteria:

* concomitantly using a strong inhibitor or inducer of CYP P450

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the University Medical Center Groningen who receive voriconazole
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Plamsa concentration of voriconazole and voriconazole N-oxide in patients during a severe inflammation | Up to 1 month
  Plasma concentrations of voriconazole and voriconazole N-oxide will be determined using a validated method involving LC-MS/MS

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Klomp SD, Veringa A, Alffenaar JC, de Boer MGJ, Span LFR, Guchelaar HJ, Swen JJ. Inflammation altered correlation between CYP2C19 genotype and CYP2C19 activity in patients receiving voriconazole. Clin Transl Sci. 2024 Jul;17(7):e13887. doi: 10.1111/cts.13887. PMID 39010708